CLINICAL TRIAL: NCT01248091
Title: The Effect of Nitroprusside on the IUD Insertion Experience in Nulliparous Women: a Pilot Study
Brief Title: The Effect of Nitroprusside on Intrauterine Device (IUD) Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Paula Bednarek, MD, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Version 1.0
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Cervical Pain; Pelvic Pain
Keywords: IUD, Insertion, Decrease, Pain
MeSH Terms: conditions — Neck Pain; Pelvic Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo gel (Placebo Comparator)
  Interventions: Procedure: Placebo Gel
- Nitroprusside Gel (Experimental)
  Interventions: Procedure: Nitroprusside Gel

INTERVENTIONS:
Procedure: Nitroprusside Gel — 10 cc nitroprusside gel
  Arms: Nitroprusside Gel
Procedure: Placebo Gel — half of the subjects will receive nitroprusside gel for IUD insertion and the other half will receive a placebo gel.
  Arms: Placebo gel

SUMMARY:
Increasing accessibility of long-acting reversible contraceptive methods, like intrauterine devices (IUDs), is an important strategy to reduce the risk of unintended pregnancy. Unfortunately, fear of IUD insertion in women who have not had children is common among health care providers and women alike, and this limits IUD use. To increase acceptance of this highly effective contraceptive, there is need to investigate novel, low cost, easily applied and accessible techniques to improve the insertion experience. This is a pilot study to evaluate the efficacy and tolerability of nitroprusside gel applied intracervically as an intervention to improve the IUD insertion experience for both patient and provider.

DETAILED DESCRIPTION:
Subjects who are have already scheduled an IUD insertion will be asked to join this study assessing whether or not nitroprusside gel helps with IUD insertion process. Only healthy, nulliparous women between the ages of 18 and 45 will be recruited. Nulliparous women report much more pain associated with IUD insertion than parous women so the possibility of being able to measure the effect of nitroprusside vs placebo is more likely. The primary outcome, pain with IUD insertion, and the secondary outcomes, such as satisfaction and provider ease of IUD insertion, will be compared between the study groups as well.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45,
* Generally Healthy.
* requesting LNG-IUS for contraception as the primary indication

Exclusion Criteria:

* previous pregnancy beyond 20 weeks,
* previous IUD placement or attempted placement,
* allergy to nitroprusside,
* history of migraines,
* history of heart disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy and tolerability of nitroprusside gel applied intracervically as an intervention to improve the IUD insertion experience for both patient and provider. | over one year

CONTACTS AND LOCATIONS:
Overall Officials: Paula Bednarek, MD MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Bednarek PH, Micks EA, Edelman AB, Li H, Jensen JT. The effect of nitroprusside on IUD insertion experience in nulliparous women: a pilot study. Contraception. 2013 Apr;87(4):421-5. doi: 10.1016/j.contraception.2012.10.030. Epub 2012 Dec 4. PMID 23218853